CLINICAL TRIAL: NCT04641221
Title: Optimization and Multi-Site Feasibility of Yoga for Chronic Pain in People in YOGAMAT-II - Phase II
Acronym: YOGAMAT-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: 202002-002-2; R01AT010863 (NIH)
Record Dates: First submitted 2020-11-16; First posted 2020-11-23 (Actual); Results first posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use; Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- No Video/No One-on-One/No Text/No Incentive (Active Comparator): This group does not receive Personal Practice Videos, or One-on-One individual sessions with a Yoga Instructor, or prompting Text messages, or financial Incentives to attend yoga classes
  Interventions: Behavioral: Weekly Yoga Classes
- No Video/No One-on-One/No Text/Yes Incentive (Active Comparator): This group does not receive Personal Practice Videos, or One-on-One individual sessions with a Yoga Instructor, or prompting Text messages, but DOES receive financial Incentives to attend yoga classes
  Interventions: Behavioral: Weekly Yoga Classes
- No Video/No One-on-One/Yes Text/No Incentive (Active Comparator): This group does not receive Personal Practice Videos, or One-on-One individual sessions with a Yoga Instructor, or financial Incentives to attend yoga classes, but DOES receive prompting Text messages
  Interventions: Behavioral: Weekly Yoga Classes
- No Video/No One-on-One/Yes Text/Yes Incentive (Active Comparator): This group does not receive Personal Practice Videos, or One-on-One individual sessions with a Yoga Instructor, but DOES receive prompting Text messages and financial Incentives to attend yoga classes
  Interventions: Behavioral: Weekly Yoga Classes
- No Video/Yes One-on-One/No Text/No Incentive (Active Comparator): This group does not receive Personal Practice Videos or prompting Text messages or financial Incentives to attend yoga classes, but DOES receive One-on-One individual sessions with a Yoga Instructor
  Interventions: Behavioral: Weekly Yoga Classes
- No Video/Yes One-on-One/No Text/Yes Incentive (Active Comparator): This group does not receive Personal Practice Videos or prompting Text messages, but DOES receive One-on-One individual sessions with a Yoga Instructor, and financial Incentives to attend yoga classes
  Interventions: Behavioral: Weekly Yoga Classes
- No Video/Yes One-on-One/Yes Text/No Incentive (Active Comparator): This group does not receive Personal Practice Videos or financial Incentives to attend yoga classes, but DOES receive One-on-One individual sessions with a Yoga Instructor and prompting Text messages
  Interventions: Behavioral: Weekly Yoga Classes
- No Video/Yes One-on-One/Yes Text/Yes Incentive (Active Comparator): This group does not receive Personal Practice Videos, but DOES receive One-on-One individual sessions with a Yoga Instructor, prompting Text messages, and financial Incentives to attend yoga classes
  Interventions: Behavioral: Weekly Yoga Classes
- Yes Video/No One-on-One/No Text/No Incentive (Active Comparator): This group does not receive One-on-One individual sessions with a Yoga Instructor, or prompting Text messages, or financial Incentives to attend yoga classes, but DOES receive Personal Practice Videos
  Interventions: Behavioral: Weekly Yoga Classes
- Yes Video/No One-on-One/No Text/Yes Incentive (Active Comparator): This group does not receive One-on-One individual sessions with a Yoga Instructor or prompting Text messages, but DOES receive Personal Practice Videos and financial Incentives to attend yoga classes
  Interventions: Behavioral: Weekly Yoga Classes
- Yes Video/No One-on-One/Yes Text/No Incentive (Active Comparator): This group does not receive One-on-One individual sessions with a Yoga Instructor or financial Incentives to attend yoga classes, but DOES receive Personal Practice Videos and prompting Text messages
  Interventions: Behavioral: Weekly Yoga Classes
- Yes Video/No One-on-One/Yes Text/Yes Incentive (Active Comparator): This group does not receive One-on-One individual sessions with a Yoga Instructor, but DOES receive Personal Practice Videos, prompting Text messages, and financial Incentives to attend yoga classes
  Interventions: Behavioral: Weekly Yoga Classes
- Yes Video/Yes One-on-One/No Text/No Incentive (Active Comparator): This group does not receive prompting Text messages or financial Incentives to attend yoga classes, but DOES receive Personal Practice Videos and One-on-One individual sessions with a Yoga Instructor
  Interventions: Behavioral: Weekly Yoga Classes
- Yes Video/Yes One-on-One/No Text/Yes Incentive (Active Comparator): This group does not receive prompting Text messages, but DOES receive Personal Practice Videos, One-on-One individual sessions with a Yoga Instructor, and financial Incentives to attend yoga classes
  Interventions: Behavioral: Weekly Yoga Classes
- Yes Video/Yes One-on-One/Yes Text/No Incentive (Active Comparator): This group does not receive financial Incentives to attend yoga classes, but DOES receive Personal Practice Videos, One-on-One individual sessions with a Yoga Instructor and prompting Text messages
  Interventions: Behavioral: Weekly Yoga Classes
- Yes Video/Yes One-on-One/Yes Text/Yes Incentive (Active Comparator): This group receives Personal Practice Videos, One-on-One individual sessions with a Yoga Instructor, prompting Text messages, and financial Incentives to attend yoga classes
  Interventions: Behavioral: Weekly Yoga Classes

INTERVENTIONS:
Behavioral: Weekly Yoga Classes — All participants are invited to attend weekly yoga classes.

SUMMARY:
Phase 2 - Multiphase Optimization Strategy (MOST) Optimization Phase:

1. To conduct a factorial experiment that will allow us to evaluate the impact of each of the 4 intervention components on yoga dosage received. We will enroll a total n=192. All participants will receive the core yoga intervention, with random assignment to the four intervention components outlined above.
2. Use results from Phase 2 to choose an efficient combination of intervention components that, together with standard yoga classes, maximizes yoga dosage.
3. Examine mechanisms by which components are hypothesized to work.

DETAILED DESCRIPTION:
In Phase 2, we will conduct a fully powered optimization trial. We will enroll 192 participants, planning to role approximately equal numbers of participants in both sites. In both phases, all participants will receive the core yoga intervention (12 weeks of weekly manualized yoga classes), with random assignment to the 4 key intervention components. Participants will be patients enrolled in methadone (MMT) or buprenorphine/naloxone (BUP) treatment with chronic pain. Enrollment period for this phase will last approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in MMT or BUP treatment for > 3 months
* Plan to continue treatment for next 6 months
* Chronic pain, defined as pain for at least half the days over the previous three months, a mean score of 4 or higher on the Brief Pain Interference Scale (BPI; with reference to chronic pain), and pain severity of 4 or higher on a Visual Analog Scale (0-10) indicating "worst pain in the last week." Pain severity score will also refer to the areas of their body in which they have chronic pain.
* Aged > 18
* Proficiency in English sufficient to engage in informed consent in English, understand classes taught in English, and read short sentences
* Available at least one of the times study classes are offered.

Exclusion Criteria:

* Currently taking yoga classes or practicing yoga at home once per week or more often.
* Medical conditions that would make participation in yoga unsafe or not possible, including active malignancy treatment, fracture, recent joint surgery, use of assistive ambulatory devices other than a cane. . (In cases where this is unclear, site PI will make final determination based on available evidence.)
* Severe or progressive neurologic deficits. (In cases where this is unclear, site PI will make final determination based on available evidence.)
* Other severe disabling chronic medical and/or psychiatric comorbidities deemed by the site PI on a case-by-case basis to prevent safe or adequate participation in the study (e.g., cognitive impairment that prevents a participant from understanding assessments; history of disruptive behavior in medical settings; severe disabling heart failure or lung disease)
* Surgery requiring overnight hospitalization planned in the next 3 months
* Pregnancy
* No access to a reasonably safe, reliable place to engage in personal yoga practice and a private space to participate in online yoga classes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Boston Medical Center, Boston, Massachusetts
  - CODAC Behavioral Healthcare, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Uebelacker LA, Braun TD, Taylor LE, Saper R, Baldwi M, Abrantes A, Tremont G, Toribio A, Kirshy S, Koch R, Lorin L, Van Noppen D, Anderson B, Roseen EJ, Stein MD. Evaluation of intervention components to maximize yoga practice among people with chronic pain taking opioid agonist therapy: A factorial experiment using the multiphase optimization strategy framework. Contemp Clin Trials. 2024 Feb;137:107411. doi: 10.1016/j.cct.2023.107411. Epub 2023 Dec 14. PMID 38103784

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For these purposes, we defined completion as completing the BPI at Month 3 or Month 12
Period: First 3 months
Arm/Group | No Video/No One-on-One/No Text/No Incentive | No Video/No One-on-One/No Text/Yes Incentive | No Video/No One-on-One/Yes Text/No Incentive | No Video/No One-on-One/Yes Text/Yes Incentive | No Video/Yes One-on-One/No Text/No Incentive | No Video/Yes One-on-One/No Text/Yes Incentive | No Video/Yes One-on-One/Yes Text/No Incentive | No Video/Yes One-on-One/Yes Text/Yes Incentive | Yes Video/No One-on-One/No Text/No Incentive | Yes Video/No One-on-One/No Text/Yes Incentive | Yes Video/No One-on-One/Yes Text/No Incentive | Yes Video/No One-on-One/Yes Text/Yes Incentive | Yes Video/Yes One-on-One/No Text/No Incentive | Yes Video/Yes One-on-One/No Text/Yes Incentive | Yes Video/Yes One-on-One/Yes Text/No Incentive | Yes Video/Yes One-on-One/Yes Text/Yes Incentive
Started | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Completed | 10 | 11 | 9 | 9 | 9 | 12 | 7 | 11 | 6 | 9 | 10 | 6 | 8 | 8 | 5 | 8
Not Completed | 2 | 1 | 3 | 3 | 3 | 0 | 5 | 1 | 6 | 3 | 2 | 6 | 4 | 4 | 7 | 4
Period: All 12 months
Arm/Group | No Video/No One-on-One/No Text/No Incentive | No Video/No One-on-One/No Text/Yes Incentive | No Video/No One-on-One/Yes Text/No Incentive | No Video/No One-on-One/Yes Text/Yes Incentive | No Video/Yes One-on-One/No Text/No Incentive | No Video/Yes One-on-One/No Text/Yes Incentive | No Video/Yes One-on-One/Yes Text/No Incentive | No Video/Yes One-on-One/Yes Text/Yes Incentive | Yes Video/No One-on-One/No Text/No Incentive | Yes Video/No One-on-One/No Text/Yes Incentive | Yes Video/No One-on-One/Yes Text/No Incentive | Yes Video/No One-on-One/Yes Text/Yes Incentive | Yes Video/Yes One-on-One/No Text/No Incentive | Yes Video/Yes One-on-One/No Text/Yes Incentive | Yes Video/Yes One-on-One/Yes Text/No Incentive | Yes Video/Yes One-on-One/Yes Text/Yes Incentive
Started | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Completed | 10 | 11 | 9 | 8 | 6 | 10 | 7 | 8 | 5 | 9 | 8 | 10 | 6 | 9 | 7 | 9
Not Completed | 2 | 1 | 3 | 4 | 6 | 2 | 5 | 4 | 7 | 3 | 4 | 2 | 6 | 3 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Video/No One-on-One/No Text/No Incentive | No Video/No One-on-One/No Text/Yes Incentive | No Video/No One-on-One/Yes Text/No Incentive | No Video/No One-on-One/Yes Text/Yes Incentive | No Video/Yes One-on-One/No Text/No Incentive | No Video/Yes One-on-One/No Text/Yes Incentive | No Video/Yes One-on-One/Yes Text/No Incentive | No Video/Yes One-on-One/Yes Text/Yes Incentive | Yes Video/No One-on-One/No Text/No Incentive | Yes Video/No One-on-One/No Text/Yes Incentive | Yes Video/No One-on-One/Yes Text/No Incentive | Yes Video/No One-on-One/Yes Text/Yes Incentive | Yes Video/Yes One-on-One/No Text/No Incentive | Yes Video/Yes One-on-One/No Text/Yes Incentive | Yes Video/Yes One-on-One/Yes Text/No Incentive | Yes Video/Yes One-on-One/Yes Text/Yes Incentive | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 192
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age in years
  Years | 44.8 (11.7) | 43.0 (8.6) | 41.8 (8.1) | 45.7 (8.9) | 43.1 (10.1) | 47.0 (13.5) | 43.8 (11.0) | 47.2 (10.4) | 42.4 (8.9) | 49.4 (10.5) | 39.9 (9.7) | 45.8 (11.2) | 43.2 (9.5) | 43.9 (10.6) | 48.0 (10.8) | 48.4 (12.0) | 44.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 7 | 9 | 11 | 6 | 6 | 8 | 10 | 6 | 10 | 8 | 10 | 5 | 7 | 8 | 124
  Male | 5 | 6 | 5 | 3 | 1 | 6 | 6 | 4 | 2 | 6 | 2 | 4 | 2 | 7 | 5 | 4 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 8
  Black or African American | 1 | 2 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 2 | 0 | 1 | 2 | 2 | 19
  White | 10 | 7 | 9 | 9 | 9 | 10 | 8 | 10 | 12 | 8 | 9 | 7 | 9 | 11 | 9 | 9 | 146
  More than one race | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 2 | 1 | 2 | 2 | 0 | 0 | 0 | 13
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 2 | 1 | 0 | 1 | 2 | 1 | 19
  Not Hispanic or Latino | 11 | 10 | 9 | 11 | 12 | 12 | 11 | 11 | 11 | 10 | 10 | 11 | 12 | 11 | 10 | 11 | 173
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Rhode Island | 3 | 2 | 6 | 7 | 4 | 7 | 4 | 4 | 5 | 5 | 6 | 5 | 5 | 5 | 3 | 5 | 76
  United States: Massachusetts | 9 | 10 | 5 | 5 | 8 | 3 | 8 | 8 | 6 | 7 | 6 | 7 | 7 | 6 | 9 | 6 | 110
  United States: Ohio | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 6
Medication for Addiction Treatment [Count of Participants; unit: Participants] — Methadone or buprenorphine
  Participants
    Methadone | 7 | 3 | 5 | 8 | 5 | 8 | 6 | 8 | 7 | 5 | 6 | 6 | 5 | 6 | 6 | 5 | 96
    Buprenorphine | 5 | 9 | 7 | 4 | 7 | 4 | 6 | 4 | 5 | 7 | 6 | 6 | 7 | 6 | 6 | 7 | 96

OUTCOME MEASURES:

1. Primary Outcome: Yoga Dosage
Description: Total minutes per week practicing yoga, including in class and outside of class, assessed weekly via interview
Time Frame: 3 months
Measure: Mean (90% Confidence Interval); unit: Total yoga Minutes
Arm/Group | No Video/No One-on-One/No Text/No Incentive | No Video/No One-on-One/No Text/Yes Incentive | No Video/No One-on-One/Yes Text/No Incentive | No Video/No One-on-One/Yes Text/Yes Incentive | No Video/Yes One-on-One/No Text/No Incentive | No Video/Yes One-on-One/No Text/Yes Incentive | No Video/Yes One-on-One/Yes Text/No Incentive | No Video/Yes One-on-One/Yes Text/Yes Incentive | Yes Video/No One-on-One/No Text/No Incentive | Yes Video/No One-on-One/No Text/Yes Incentive | Yes Video/No One-on-One/Yes Text/No Incentive | Yes Video/No One-on-One/Yes Text/Yes Incentive | Yes Video/Yes One-on-One/No Text/No Incentive | Yes Video/Yes One-on-One/No Text/Yes Incentive | Yes Video/Yes One-on-One/Yes Text/No Incentive | Yes Video/Yes One-on-One/Yes Text/Yes Incentive
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Total yoga Minutes | 164.5 [100.2 to 228.8] | 99.4 [67.4 to 131.5] | 139.1 [108.8 to 169.4] | 102.2 [72.2 to 132.1] | 116.6 [73.9 to 159.3] | 154.8 [113.8 to 195.8] | 84.5 [68.5 to 100.6] | 185.6 [118.9 to 252.4] | 89.7 [72.6 to 106.8] | 90.9 [68.5 to 113.4] | 111.4 [67.0 to 155.7] | 122.3 [98.1 to 146.4] | 145.8 [99.6 to 192.0] | 144.9 [116.6 to 173.1] | 167.0 [129.1 to 204.8] | 117.2 [83.0 to 151.4]
Statistical Analysis 1: Comparison: No Video/No One-on-One/No Text/No Incentive vs No Video/No One-on-One/No Text/Yes Incentive vs No Video/No One-on-One/Yes Text/No Incentive vs No Video/No One-on-One/Yes Text/Yes Incentive vs No Video/Yes One-on-One/No Text/No Incentive vs No Video/Yes One-on-One/No Text/Yes Incentive vs No Video/Yes One-on-One/Yes Text/No Incentive vs No Video/Yes One-on-One/Yes Text/Yes Incentive vs Yes Video/No One-on-One/No Text/No Incentive vs Yes Video/No One-on-One/No Text/Yes Incentive vs Yes Video/No One-on-One/Yes Text/No Incentive vs Yes Video/No One-on-One/Yes Text/Yes Incentive vs Yes Video/Yes One-on-One/No Text/No Incentive vs Yes Video/Yes One-on-One/No Text/Yes Incentive vs Yes Video/Yes One-on-One/Yes Text/No Incentive vs Yes Video/Yes One-on-One/Yes Text/Yes Incentive; There were four potential intervention components. This study used a 2x2x2x2 factorial design. Thus, we analyzed main and interaction effects for the four potential intervention components; Test type: Superiority; p = 0.028, zero-inflated negative-binomial (ZINB) — main effect for one-on-one sessions; We specified a multilevel (week nested within participant) model which included terms for each main effect and each interaction effect and covariates; incidence rate ratio = 1.10, 90% CI 2-sided [1.02 to 1.18] — Main effect for One-one sessions
Statistical Analysis 2: Comparison: No Video/No One-on-One/No Text/No Incentive vs No Video/No One-on-One/No Text/Yes Incentive vs No Video/No One-on-One/Yes Text/No Incentive vs No Video/No One-on-One/Yes Text/Yes Incentive vs No Video/Yes One-on-One/No Text/No Incentive vs No Video/Yes One-on-One/No Text/Yes Incentive vs No Video/Yes One-on-One/Yes Text/No Incentive vs No Video/Yes One-on-One/Yes Text/Yes Incentive vs Yes Video/No One-on-One/No Text/No Incentive vs Yes Video/No One-on-One/No Text/Yes Incentive vs Yes Video/No One-on-One/Yes Text/No Incentive vs Yes Video/No One-on-One/Yes Text/Yes Incentive vs Yes Video/Yes One-on-One/No Text/No Incentive vs Yes Video/Yes One-on-One/No Text/Yes Incentive vs Yes Video/Yes One-on-One/Yes Text/No Incentive vs Yes Video/Yes One-on-One/Yes Text/Yes Incentive; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Interaction effect for one-on-one sessions and incentives for participation; p = 0.039, zero-inflated negative binomial; incidence rate ratio = 1.09, 90% CI 2-sided [1.02 to 1.17] — Interaction effect for one-on-one sessions and incentives for participation
Statistical Analysis 3: Comparison: No Video/No One-on-One/No Text/No Incentive vs No Video/No One-on-One/No Text/Yes Incentive vs No Video/No One-on-One/Yes Text/No Incentive vs No Video/No One-on-One/Yes Text/Yes Incentive vs No Video/Yes One-on-One/No Text/No Incentive vs No Video/Yes One-on-One/No Text/Yes Incentive vs No Video/Yes One-on-One/Yes Text/No Incentive vs No Video/Yes One-on-One/Yes Text/Yes Incentive vs Yes Video/No One-on-One/No Text/No Incentive vs Yes Video/No One-on-One/No Text/Yes Incentive vs Yes Video/No One-on-One/Yes Text/No Incentive vs Yes Video/No One-on-One/Yes Text/Yes Incentive vs Yes Video/Yes One-on-One/No Text/No Incentive vs Yes Video/Yes One-on-One/No Text/Yes Incentive vs Yes Video/Yes One-on-One/Yes Text/No Incentive vs Yes Video/Yes One-on-One/Yes Text/Yes Incentive; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.001, Zero-inflated negative binomial — 3-way interaction: study videos X one-on-one X incentives for class attendance; incident rate ratio = 0.86, 90% CI 2-sided [0.80 to 0.93] — 3-way interaction: study videos X one-on-one X incentives for class attendance

ADVERSE EVENTS:
Time Frame: 12 months
Description: We inquired about adverse events at 3 months, 6 months, and 12 months.
Arm/Group | No Video/No One-on-One/No Text/No Incentive | No Video/No One-on-One/No Text/Yes Incentive | No Video/No One-on-One/Yes Text/No Incentive | No Video/No One-on-One/Yes Text/Yes Incentive | No Video/Yes One-on-One/No Text/No Incentive | No Video/Yes One-on-One/No Text/Yes Incentive | No Video/Yes One-on-One/Yes Text/No Incentive | No Video/Yes One-on-One/Yes Text/Yes Incentive | Yes Video/No One-on-One/No Text/No Incentive | Yes Video/No One-on-One/No Text/Yes Incentive | Yes Video/No One-on-One/Yes Text/No Incentive | Yes Video/No One-on-One/Yes Text/Yes Incentive | Yes Video/Yes One-on-One/No Text/No Incentive | Yes Video/Yes One-on-One/No Text/Yes Incentive | Yes Video/Yes One-on-One/Yes Text/No Incentive | Yes Video/Yes One-on-One/Yes Text/Yes Incentive
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 4/12 | 3/12 | 3/12 | 2/12 | 3/12 | 1/12 | 2/12 | 1/12 | 2/12 | 1/12 | 2/12 | 4/12 | 1/12 | 1/12 | 3/12 | 1/12
Other Adverse Events (participants affected / at risk) | 9/12 | 9/12 | 6/12 | 7/12 | 5/12 | 8/12 | 10/12 | 5/12 | 8/12 | 9/12 | 7/12 | 8/12 | 8/12 | 6/12 | 7/12 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Video/No One-on-One/No Text/No Incentive (N=12) | No Video/No One-on-One/No Text/Yes Incentive (N=12) | No Video/No One-on-One/Yes Text/No Incentive (N=12) | No Video/No One-on-One/Yes Text/Yes Incentive (N=12) | No Video/Yes One-on-One/No Text/No Incentive (N=12) | No Video/Yes One-on-One/No Text/Yes Incentive (N=12) | No Video/Yes One-on-One/Yes Text/No Incentive (N=12) | No Video/Yes One-on-One/Yes Text/Yes Incentive (N=12) | Yes Video/No One-on-One/No Text/No Incentive (N=12) | Yes Video/No One-on-One/No Text/Yes Incentive (N=12) | Yes Video/No One-on-One/Yes Text/No Incentive (N=12) | Yes Video/No One-on-One/Yes Text/Yes Incentive (N=12) | Yes Video/Yes One-on-One/No Text/No Incentive (N=12) | Yes Video/Yes One-on-One/No Text/Yes Incentive (N=12) | Yes Video/Yes One-on-One/Yes Text/No Incentive (N=12) | Yes Video/Yes One-on-One/Yes Text/Yes Incentive (N=12)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flu-like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders - Other, specify (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychiatric Disorders- Other, Specify (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Social circumstances - Other, specify (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Video/No One-on-One/No Text/No Incentive (N=12) | No Video/No One-on-One/No Text/Yes Incentive (N=12) | No Video/No One-on-One/Yes Text/No Incentive (N=12) | No Video/No One-on-One/Yes Text/Yes Incentive (N=12) | No Video/Yes One-on-One/No Text/No Incentive (N=12) | No Video/Yes One-on-One/No Text/Yes Incentive (N=12) | No Video/Yes One-on-One/Yes Text/No Incentive (N=12) | No Video/Yes One-on-One/Yes Text/Yes Incentive (N=12) | Yes Video/No One-on-One/No Text/No Incentive (N=12) | Yes Video/No One-on-One/No Text/Yes Incentive (N=12) | Yes Video/No One-on-One/Yes Text/No Incentive (N=12) | Yes Video/No One-on-One/Yes Text/Yes Incentive (N=12) | Yes Video/Yes One-on-One/No Text/No Incentive (N=12) | Yes Video/Yes One-on-One/No Text/Yes Incentive (N=12) | Yes Video/Yes One-on-One/Yes Text/No Incentive (N=12) | Yes Video/Yes One-on-One/Yes Text/Yes Incentive (N=12)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (5) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5) | 2 (2) | 3 (4) | 4 (7) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 2 (3) | 0 (0) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (5) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flu-like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Flu-like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders - Other, specify (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders - Other, specify (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Psychiatric Disorders- Other, Specify (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT04641221/Prot_SAP_000.pdf